CLINICAL TRIAL: NCT00777634
Title: Follow-Up Extension to the Family Study of Binge Eating Disorder
Status: Completed | Type: Observational
Sponsor: Mclean Hospital (Other)
Collaborators: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, James I. Hudson, MD, Professor of Psychiatry, Harvard Medical School, Mclean Hospital
Other Study IDs: 2005-P-000779
Record Dates: First submitted 2008-10-20; First posted 2008-10-22 (Estimated); Results first posted 2012-05-29 (Estimated); Last update posted 2012-05-29 (Estimated); Status verified 2012-04

CONDITIONS: Binge Eating Disorder
Keywords: Binge Eating Disorder; Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Binge eating disorder (BED): Individuals who meet criteria for binge eating disorder.
  Interventions: Other: No intervention.
- Without BED: Individuals who do not meet criteria for binge eating disorder.
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention. — There is no intervention used in this study. Cohort members are interviewed and blood pressure, weight, and laboratory specimens are obtained.

SUMMARY:
This study involves a 2.5 and 5 year follow-up interview for individuals who participated in the initial family study of binge eating disorder. The study includes individuals with and without eating disorder as well as their first degree relatives. As part of the study, participants will be interviewed about their current psychiatric and medical symptoms, their blood pressure will be measured, and laboratory specimens will be obtained.

DETAILED DESCRIPTION:
Previously we completed a family interview study of 150 individuals with binge eating disorder, 150 matched controls, and approximately 888 of their first degree relatives. In follow-up to this, we are interviewing these individuals again at 2.5 and 5 years after their initial interview. During the course of the interview, individuals are asked about their psychiatric and medical history and blood pressure and laboratory specimens are obtained to measure, among other things, fasting lipids and glucose.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with or without binge eating disorder and their family members who participated in the initial family study of binge eating disorder and agree to be followed up at 2.5 and 5 years.

Exclusion Criteria:

* Unwilling or unable to participate in the follow-up study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study includes individuals with binge eating disorder, individuals without binge eating disorder, and their relatives.
Sampling Method: Non-Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2005-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James I Hudson, M.D., Sc.D., Principal Investigator — Mclean Hospital; Harrison G Pope, M.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

REFERENCES:
- [Derived] Hudson JI, Lalonde JK, Coit CE, Tsuang MT, McElroy SL, Crow SJ, Bulik CM, Hudson MS, Yanovski JA, Rosenthal NR, Pope HG Jr. Longitudinal study of the diagnosis of components of the metabolic syndrome in individuals with binge-eating disorder. Am J Clin Nutr. 2010 Jun;91(6):1568-73. doi: 10.3945/ajcn.2010.29203. Epub 2010 Apr 28. PMID 20427731

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Binge Eating Disorder (BED) | Without BED
Started | 134 | 134
Completed | 129 | 133
Not Completed | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Binge Eating Disorder (BED) | Without BED | Total
Number analyzed (Participants) | 134 | 134 | 268
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 134 | 134 | 268
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 47.0 (13.2) | 47.8 (12.9) | 47.4 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 102 | 209
  Male | 27 | 32 | 59
Region of Enrollment [Number; unit: participants]
  United States | 134 | 134 | 268

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Diagnosis of Dyslipidemia
Description: The number of participants to acquire a new diagnosis of high cholesterol (dyslipidemia) over the course of the baseline to five-year followup.
Time Frame: Baseline to 5 years
Measure: Number; unit: participants
Arm/Group | Binge Eating Disorder (BED) | Without BED
Number analyzed (Participants) | 129 | 133
participants | 34 | 18

2. Primary Outcome: Incidence of Diagnosis of Hypertension
Description: The number of participants to acquire a new diagnosis of high blood pressure(hypertension) over the course of the baseline to five-year followup.
Time Frame: Baseline to 5 years
Measure: Number; unit: participants
Arm/Group | Binge Eating Disorder (BED) | Without BED
Number analyzed (Participants) | 129 | 133
participants | 25 | 18

3. Primary Outcome: Incidence of Diagnosis of Type 2 Diabetes
Description: The number of participants to acquire a new diagnosis of Type 2 Diabetes over the course of the baseline to five-year followup.
Time Frame: Baseline to 5 years
Measure: Number; unit: participants
Arm/Group | Binge Eating Disorder (BED) | Without BED
Number analyzed (Participants) | 129 | 133
participants | 13 | 10

4. Primary Outcome: Incidence of Diagnosis of Any Metabolic Syndrome Component
Description: The number of participants to acquire a new diagnosis of one component of metabolic syndrome. Metabolic syndrome can include abdominal obesity, high blood pressure, high cholesterol, etc.
Time Frame: Baseline to 5 years
Measure: Number; unit: participants
Arm/Group | Binge Eating Disorder (BED) | Without BED
Number analyzed (Participants) | 129 | 133
participants | 53 | 37

5. Primary Outcome: Incidence of Diagnosis of Two or More Metabolic Syndrome Components
Description: The number of participants to acquire a new diagnosis of two or more components of metabolic syndrome. Metabolic syndrome can include abdominal obesity, high blood pressure, high cholesterol, etc.
Time Frame: Baseline to 5 years
Measure: Number; unit: participants
Arm/Group | Binge Eating Disorder (BED) | Without BED
Number analyzed (Participants) | 129 | 133
participants | 18 | 8

6. Primary Outcome: Incidence of Diagnosis of Three or More Metabolic Syndrome Components
Description: The number of participants to acquire a new diagnosis of three or more components of metabolic syndrome. Metabolic syndrome can include abdominal obesity, high blood pressure, high cholesterol, etc.
Time Frame: Baseline to 5 years
Measure: Number; unit: participants
Arm/Group | Binge Eating Disorder (BED) | Without BED
Number analyzed (Participants) | 129 | 133
participants | 1 | 1

ADVERSE EVENTS:
Description: This was an observational study, and so no participants were at risk. No intervention was administered.
Arm/Group | Binge Eating Disorder (BED) | Without BED
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No